CLINICAL TRIAL: NCT03712670
Title: Treatment of Exudative Age-Related Macular Degeneration With Aflibercept Combined With Pranoprofen Eye Drops or Nutraceutical Support With Omega-3: A Randomized Trial
Brief Title: Nutraceutical Support With Omega-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Francesco Semeraro, Dr. Francesco Semeraro, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oral001
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases | interventions — aflibercept; pyranoprofen; Carotenoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AM group (Active Comparator): Intravitreal aflibercept monotherapy
  Interventions: Drug: Aflibercept
- AP group (Experimental): Intravitreal aflibercept along with 0.1% pranoprofen
  Interventions: Drug: Aflibercept; Drug: Pranoprofen
- AN group (Experimental): Intravitreal aflibercept plus daily supplementation of nutraceutical tablets
  Interventions: Drug: Aflibercept; Dietary Supplement: Carotenoids

INTERVENTIONS:
Drug: Aflibercept — monthly intravitreal injections
Drug: Pranoprofen — 0.1% pranoprofen 3 times a day topical eye drops administration
  Arms: AP group
Dietary Supplement: Carotenoids — daily supplementation of nutraceutical tablets containing the AREDS2 formulation
  Arms: AN group

SUMMARY:
Although evidence have clearly proved that intravitreal injection of vascular endothelial growth factor antagonists prevents vision loss and may even improve visual acuity in patients with neovascular AMD, a significant percentage of patients continue to lose visual acuity. Moreover, monthly intravitreal injections represent a burden for society as well as the caregiver.

Combination therapy with either topical 0.1% pranoprofen or nutraceutical support with AREDS2 formula plus omega-3 might act synergistically with intravitreal injection, offering valuable therapeutic support to aflibercept injections in patients requiring long-term treatment.

ELIGIBILITY:
Inclusion Criteria:

* provision of written informed consent and compliance with study assessments for the full duration of the study
* age > 40 years
* presence of treatment-naïve neovascular AMD

Exclusion Criteria:

* any previous intravitreal treatment
* previous laser treatment in the study eye
* myopia > 7 diopters in the study eye
* concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy and advanced glaucoma)
* concurrent corneal epithelial disruption or any condition that would affect the ability of the cornea to heal
* known sensitivity to any component of the formulations being investigated.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Central Retinal Thickness (microns) | 12-month
  Optical Coherence Tomography will be used to assess central retinal thickness.
Visual Acuity (LogMAR) | 12-month
  ETDRS charts will be used to assess best corrected visual acuity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AREDS2 Research Group; Chew EY, Clemons T, SanGiovanni JP, Danis R, Domalpally A, McBee W, Sperduto R, Ferris FL. The Age-Related Eye Disease Study 2 (AREDS2): study design and baseline characteristics (AREDS2 report number 1). Ophthalmology. 2012 Nov;119(11):2282-9. doi: 10.1016/j.ophtha.2012.05.027. Epub 2012 Jul 26. PMID 22840421
- [Background] Age-Related Eye Disease Study 2 (AREDS2) Research Group; Chew EY, Clemons TE, Sangiovanni JP, Danis RP, Ferris FL 3rd, Elman MJ, Antoszyk AN, Ruby AJ, Orth D, Bressler SB, Fish GE, Hubbard GB, Klein ML, Chandra SR, Blodi BA, Domalpally A, Friberg T, Wong WT, Rosenfeld PJ, Agron E, Toth CA, Bernstein PS, Sperduto RD. Secondary analyses of the effects of lutein/zeaxanthin on age-related macular degeneration progression: AREDS2 report No. 3. JAMA Ophthalmol. 2014 Feb;132(2):142-9. doi: 10.1001/jamaophthalmol.2013.7376. PMID 24310343